CLINICAL TRIAL: NCT05168865
Title: Letrozole Versus Hormonal Preparation in Frozen Cycles of PCOS Patients. Randomized Controlled Study
Brief Title: Letrozole Versus Hormonal Preparation in Frozen Cycles of PCOS Patients.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unexpected slow recruitment and change of center frozen embryo transfer protocol
Sponsor: Dubai Fertility Center (Other)
Responsible Party: Principal Investigator, Mohamed Elkalyoubi, Principal investigator, Dubai Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSREC-09/2020_16
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Frozen Embryo Transfer; Polycystic Ovarian Disease; Letrozole; Hormone Replacement Therapy; Live Birth; Miscarriage
MeSH Terms: conditions — Polycystic Ovary Syndrome; Abortion, Spontaneous | interventions — Letrozole; Estradiol; Progesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS women will receive letrozole ovarian stimulation. (Experimental): Polycystic ovarian disease (PCOS) women undergoing frozen embryo transfer (FER) will use Letrozole 5 mg starting on day 3 of spontaneous menstrual period or after progesterone withdrawal bleeding for five consecutive days.
  Interventions: Drug: Letrozole 2.5mg
- PCOS women will receive Estradiol and Progesterone (hormonal endometrial preparation). (Active Comparator): PCOS women will use daily Cetorelix acetate 0.25 mg injections for 5 days from day 1-3 of the menstrual follow or after progesterone (P4) withdrawal bleeding. They will commence daily oral Estradiol Valerate (E2) 2 mg twice daily for 5 days starting from day 3 of the menstrual flow or after P4 withdrawal bleeding, then-after three times daily. When endometrial thickness reaches 7 mm or more, the dose of E2 will be reduced to 4 mg/ day. Women will start using vaginal micronized P4 100 mg three times daily starting from 8PM. After 48 hours of starting the vaginal P4, oral Dydrogesterone 10 mg three times daily will commence.
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Letrozole 2.5mg — Letrozole 5 mg starting on day 3 of spontaneous menstrual period or after progesterone withdrawal bleeding for five consecutive days.
  Other Names: estradiol and progesterone

SUMMARY:
One of the indications of freezing is to reduce the risk of ovarian hyperstimulation syndrome particularly in polycystic ovarian disease (PCOS) women. Very few RCTs addressed the issue of optimizing the endometrium for a frozen cycle. Interestingly, Letrozole for ovarian stimulation showed significantly better reproductive outcome when compared with hormone replacement therapy (HRT) cycle. In addition, HRT cycle has been associated with higher miscarriage rate when compared with natural cycle frozen embryo transfer. Nevertheless, there is not yet a well-designed prospective randomized study comparing letrozole and HRT in PCOS women undergoing frozen embryo transfer.

DETAILED DESCRIPTION:
Freezing oocytes and embryos has become an integral part of the daily IVF practice. One of the indications of freezing is to reduce the risk of ovarian hyperstimulation syndrome particularly in polycystic ovarian disease (PCOS) women.

Very few randomized control trials addressed the issue of optimizing the endometrium for a frozen cycle. As PCOS women do not regularly ovulate, most of their frozen cycles are conducted after hormonal replacement therapy (HRT) preparation of the endometrium or after ovulation induction. In HRT cycle the endometrium is prepared using exogenous estradiol and progesterone. While HRT cycles requires less monitoring and easy scheduling, it is costly, associated with increased risk of thrombosis and women must continue using the exogenous hormones up to 10 to 12 weeks of gestation.

Interestingly, Letrozole for ovarian stimulation showed significantly better reproductive outcome when compared with HRT cycles. In agreement with the previous Chinese study, a retrospective Japanese ART registry data that included 110 722 frozen cycles confirmed the superiority of letrozole. Nevertheless, there is not yet a well-designed prospective randomized study.

In addition, HRT cycle has been associated with higher miscarriage rate when compared with natural cycle frozen embryo transfer. HRT is usually used in patients with PCOS. A retrospective study including 2664 PCOS patients showed significant decrease in the pregnancy loss when letrozole was used when compared with HRT in frozen cycles.

Investigators thought of comparing letrozole and HRT in women with PCOS who are undergoing frozen cycles in PCOS women. Live birth and miscarriage rates will be the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS diagnosed with Rotterdam criteria.
* Age between 20 to 40-year-old
* Undergoing frozen oocytes intracytoplasmic sperm injection transfer or frozen embryo transfer
* Willingly accept to participate in the study

Exclusion Criteria:

* Women > 40 years old or younger than 20.
* Uterine pathology that decreases the chance of pregnancy or increases risk of miscarriage such as

  * Uterine fibroids (sub-mucous of any size or intramural of > 3 cm)
  * Uncontrolled endocrinal-pathological disease like

    * Cushing syndrome,
    * Adrenal hyperplasia,
    * Hyperprolactinemia,
    * Acromegaly,
    * Thyroid disease,
    * Diabetes mellitus, and
    * Immune disorders.
* Presence of Hydrosalpinx
* Not willing or able to sign the consent form.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
livebirth rate per embryo transfer | 9 months
  A birth after 24 weeks gestation with a baby showing signs of life.

SECONDARY OUTCOMES:
miscarriage rate per embryo transfer | 6 months
  loss of pregnancy before 24 weeks gestation
ongoing pregnancy per embryo transfer | 3 months
  ongoing viable pregnancy (by ultrasound examination at 12 weeks' gestation)